CLINICAL TRIAL: NCT00704145
Title: A Prospective Optical Coherence Tomography Study on Completeness of Strut Coverage and Vessel Wall Response at 3-6 and 9 Months Following Paclitaxel Eluting Stent Implantation in Multivessel Coronary Artery Disease
Brief Title: Optical Coherence Tomography Following Paclitaxel Eluting Stent Implantation in Multivessel Coronary Artery Disease
Acronym: OCTAXUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Collaborators: Case Western Reserve University (Other); Boston Scientific Corporation (Industry)
Responsible Party: Giulio Guagliumi, Ospedali Riuniti di Bergamo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1087/2007
Record Dates: First submitted 2008-06-20; First posted 2008-06-24 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2010-02

CONDITIONS: Coronary Artery Disease
Keywords: Drug Eluting Stents; Percutaneous Coronary Interventions; Optical Coherence Tomography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Device, paclitaxel drug-eluting stent
  Interventions: Device: Taxus Libertè™ paclitaxel drug-eluting stent

INTERVENTIONS:
Device: Taxus Libertè™ paclitaxel drug-eluting stent — device:Taxus Libertè™ (Boston Scientific,Natick,MS)assessed at different time points after implant
  Other Names: Taxus Libertè™ (Boston Scientific,Natick,MS)

SUMMARY:
A prospective Optical Coherence Tomography (OCT) study on the completeness of strut coverage and vessel wall response, at different time points (3-6-9 Months), following TAXUS Liberte stent implantation (staged procedures) in patients with multi vessel native coronary artery lesions

DETAILED DESCRIPTION:
Major concerns were addressed to the delayed healing process of drug-eluting stents in off-label indications. To date no studies have detailed the in-vivo completeness of DES coverage at different time points. The objective of this prospective study is to measure the completeness of strut coverage and vessel wall response (neointima disomogeneity, acquired late incomplete strut apposition) at different time points following paclitaxel-eluting stent implantation, in patients with multivessel disease treated with staged PCI procedures. Optical Coherence Tomography (OCT) that detects smaller degrees of stent strut coverage more accurately than IVUS will be used at different time point. Intravascular ultrasound (IVUS) will be performed as per normal practice at any index procedures and 9 months elective follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Multivessel coronary artery disease (two or 3 VD) to be treated at 2 sequences (staged procedures) with paclitaxel-polymer eluting stents
2. Native coronary artery disease with >= 75% diameter stenosis
3. Vessel size in between 2.5 and 3.5 mm.
4. Written informed consent signed

Exclusion Criteria:

1. No suitable anatomy for OCT scan: (truly ostial , tortuous anatomy, very distal lesions or vessels larger than 3.75 in reference diameter).
2. significant left main coronary artery disease,
3. lesions in bypass grafts,
4. acute myocardial infarction,
5. poor cardiac function as defined by left ventricular ejection fraction ≤ 30%.
6. allergy to aspirin and or clopidogrel/ticlopidine,
7. Renal failure with creatinine value > 2.5 mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-08 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Proportion of uncovered and/or malapposed Taxus Libertè struts at different time point after the implant, as measured by OCT | 3-6-9 months

SECONDARY OUTCOMES:
% Incomplete apposition at different point of FU (3-6-9 months) | 3-6-9 months
Proportion of neointima disomogeneity around struts at different point of FU (3-6-9 months) | 3-6-9 months
OCT Neointima thickness overtime | 3-6-9 months
Ischemia Driven Target Vessel Failure (ID-TVF) rate at 12 months | 12 months
Adjudicated MACE rate at 30 days and 12 months | 30 days and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Guagliumi, MD, Principal Investigator — Cardiovascular Department Ospedali Riuniti di Bergamo
Locations (1):
- Ospedali Riuniti di Bergamo, Bergamo, Italy

REFERENCES:
- [Background] Finn AV, Nakazawa G, Joner M, Kolodgie FD, Mont EK, Gold HK, Virmani R. Vascular responses to drug eluting stents: importance of delayed healing. Arterioscler Thromb Vasc Biol. 2007 Jul;27(7):1500-10. doi: 10.1161/ATVBAHA.107.144220. Epub 2007 May 17. PMID 17510464
- [Background] Finn AV, Joner M, Nakazawa G, Kolodgie F, Newell J, John MC, Gold HK, Virmani R. Pathological correlates of late drug-eluting stent thrombosis: strut coverage as a marker of endothelialization. Circulation. 2007 May 8;115(18):2435-41. doi: 10.1161/CIRCULATIONAHA.107.693739. Epub 2007 Apr 16. PMID 17438147
- [Background] Park DW, Yun SC, Lee SW, Kim YH, Lee CW, Hong MK, Kim JJ, Choo SJ, Song H, Chung CH, Lee JW, Park SW, Park SJ. Long-term mortality after percutaneous coronary intervention with drug-eluting stent implantation versus coronary artery bypass surgery for the treatment of multivessel coronary artery disease. Circulation. 2008 Apr 22;117(16):2079-86. doi: 10.1161/CIRCULATIONAHA.107.750109. Epub 2008 Apr 14. PMID 18413495
- [Background] Briguori C, Colombo A, Airoldi F, Focaccio A, Iakovou I, Chieffo A, Michev I, Montorfano M, Bonizzoni E, Ricciardelli B, Condorelli G. Sirolimus-eluting stent implantation in diabetic patients with multivessel coronary artery disease. Am Heart J. 2005 Oct;150(4):807-13. doi: 10.1016/j.ahj.2004.12.012. PMID 16209986
- [Background] Rodriguez AE, Mieres J, Fernandez-Pereira C, Vigo CF, Rodriguez-Alemparte M, Berrocal D, Grinfeld L, Palacios I. Coronary stent thrombosis in the current drug-eluting stent era: insights from the ERACI III trial. J Am Coll Cardiol. 2006 Jan 3;47(1):205-7. doi: 10.1016/j.jacc.2005.10.016. Epub 2005 Dec 9. No abstract available. PMID 16386687
- [Background] Matsumoto D, Shite J, Shinke T, Otake H, Tanino Y, Ogasawara D, Sawada T, Paredes OL, Hirata K, Yokoyama M. Neointimal coverage of sirolimus-eluting stents at 6-month follow-up: evaluated by optical coherence tomography. Eur Heart J. 2007 Apr;28(8):961-7. doi: 10.1093/eurheartj/ehl413. Epub 2006 Nov 29. PMID 17135281
- [Background] Takano M, Inami S, Jang IK, Yamamoto M, Murakami D, Seimiya K, Ohba T, Mizuno K. Evaluation by optical coherence tomography of neointimal coverage of sirolimus-eluting stent three months after implantation. Am J Cardiol. 2007 Apr 15;99(8):1033-8. doi: 10.1016/j.amjcard.2006.11.068. Epub 2007 Feb 23. PMID 17437723
- [Background] Yamaguchi T, Terashima M, Akasaka T, Hayashi T, Mizuno K, Muramatsu T, Nakamura M, Nakamura S, Saito S, Takano M, Takayama T, Yoshikawa J, Suzuki T. Safety and feasibility of an intravascular optical coherence tomography image wire system in the clinical setting. Am J Cardiol. 2008 Mar 1;101(5):562-7. doi: 10.1016/j.amjcard.2007.09.116. Epub 2008 Jan 10. PMID 18307999
- [Derived] Guagliumi G, Bezerra HG, Sirbu V, Ikejima H, Musumeci G, Biondi-Zoccai G, Lortkipanidze N, Fiocca L, Capodanno D, Wang W, Tahara S, Vassileva A, Matiashvili A, Valsecchi O, Costa MA. Serial assessment of coronary artery response to paclitaxel-eluting stents using optical coherence tomography. Circ Cardiovasc Interv. 2012 Feb 1;5(1):30-8. doi: 10.1161/CIRCINTERVENTIONS.111.965582. Epub 2012 Jan 31. PMID 22298797